CLINICAL TRIAL: NCT02614534
Title: Multicentre, Randomized Clinical Trial to Evaluate Safety and Efficacy of Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) With Mitomycin C Used During Surgery for Treatment of Locally Advanced Colorectal Carcinoma
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) With Mitomycin C Used During Surgery for Treatment of Locally Advanced Colorectal Carcinoma
Acronym: HIPECT4
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCO-HIP-2015-01
Record Dates: First submitted 2015-11-09; First posted 2015-11-25 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
Keywords: HIPEC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proactive cytoreductive surgery + HIPEC (Experimental): Tumoral cytoreductive surgery + apendicectomy + total omentectomy + round hepatic ligament + oophorectomy (postmenopausian women) plus HIPEC (Mytomicin C - 60 minutes).
  Interventions: Drug: MITOMYCIN-C 30 mg
- Proactive cytoreductive surgery (Active Comparator): Tumoral cytoreductive surgery + apendicectomy + total omentectomy + round hepatic ligament + oophorectomy (postmenopausian women).
  Interventions: Procedure: Proactive cytoreductive surgery

INTERVENTIONS:
Drug: MITOMYCIN-C 30 mg — Proactive cytoreductive surgery: Tumoral cytoreductive surgery + apendicectomy + total omentectomy + round hepatic ligament + oophorectomy (postmenopausian women) plus HIPEC with Mytomicin C for 60 minutes.
  Arms: Proactive cytoreductive surgery + HIPEC
Procedure: Proactive cytoreductive surgery — Proactive cytoreductive surgery: Tumoral cytoreductive surgery + apendicectomy + total omentectomy + round hepatic ligament + oophorectomy (postmenopausian women)
  Arms: Proactive cytoreductive surgery

SUMMARY:
The purpose of this study is to determine whether Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) with Mitomycin C used during surgery for treatment of locally advanced colorectal carcinoma is effective in the treatment of locally advanced colorectal carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) with Mitomycin C used during surgery for treatment of locally advanced colorectal carcinoma is effective in the treatment of locally advanced colorectal carcinoma.

The Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) is expected to be an effective treatment with minimal side effects, it has already provided clear benefits in terms of overall survival in patients with advanced cancer.

This is an attractive option for the healthcare professionals who face daily to peritoneal recurrence after performing complex surgeries, however its application is difficult due to the cost and resources increase. This leads to the necessity of administering the treatment within a clinical trials and in order to obtain a significant power this clinical trials will be multicenter and it will be performed in several Oncological surgery Units highly specialised and with extensive experience in colorectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 and 75 years;
2. Adenocarcinoma of the colon, sigma and colon-sigma joint which represent cT4a/b in line with The American Joint Committee on Cancer: the 7th edition of the AJCC cancer staging manual;
3. Lymph node involvement: N0, the presence of N1/2 according to the 7th edition of the AJCC is allowed, provided that they can be resectable;
4. Metastatic extent: M0;
5. Karnofsky index >70 or Performance status ≤2;
6. Informed consent properly completed.

Exclusion Criteria:

1. Presence of metastases (M1), in case of liver or peritoneal metastases at the time of surgery, the patient will be excluded from the trial and treated according to their new stage.
2. Presence of unresectability criteria;
3. Urgent intervention due to obstruction or perforation if there is tumor removal, prior interventions will be accepted as referrals without primary tumor removal or drainage of collections prior to scheduled surgery.
4. Extraperitoneal rectal cáncer (avoiding alterations for neoadyuvance);
5. Coexistence of another malignant neoplastic disease (synchronous tumors of the colon and upper rectum are accepted as long as the stage is equal to or less than the treated tumor).
6. Severely altered liver, kidney and cardiovascular function;
7. Intolerance to treatment;
8. Administration of chemotherapy before the trial (use of neoadyuvance is discarded);
9. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11-16 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Locoregional Control (LC) | 3 years
  Time elapsed from the surgical intervention clinical up to the date the patient is free of clinical and radiological locoregional recurrence

SECONDARY OUTCOMES:
Overall survival | 12 months and 36 months after surgery
  Evaluate the effect of the addition of HIPEC with Mitomycin C to cytoreductive surgery in 12 months and 3 years overall survival rate (%OS).
Disease Free Survival | 12 months and 36 months after surgery
  Evaluate the effect of addition of HIPEC with Mitomycin C to cytoreductive surgery in 12 months and 3 years disease free survival rate (% DFS).
Evaluation of the morbidity and mortality related with the treatment | 36 months after surgery
  Evaluate the safety (treatment-related morbidity and mortality) of addition of HIPEC with Mitomycin C to cytoreductive surgery in locally advanced colo-rectal cancer. It will be measured by the incidence rate of adverse events and deaths.
HIPEC technique operating time | 36 months after surgery
  Average operating time calculation.
HIPEC technique length of hospital stay | 36 months after surgery
  Average length of hospital stay calculation.
HIPEC technique re-admission rate | 36 months after surgery
  Average re-admission rate calculation.
HIPEC technique laparoscopic vs laparotomy approach | 36 months after surgery
  With this outcome it will be calculated the frequency of both surgery techniques and if it has any impact on the locoregional control of the disease.
HIPEC technique open vs. closed HIPEC technique | 36 months after surgery
  With this outcome it will be calculated the frequency of both surgery techniques and if it has any impact on the locoregional control of the disease.
Quality of life questionnaire QLQ-C30 | At baseline, 1 month after surgery, 6 months after surgery, 12 months after surgery, 24 months after surgery and 36 months after surgery
  With this outcome it will be calculated the effect on the quality of life of patients using questionnaire QLQ-C30.
Quality of life questionnaires QLQ-CR29 | At baseline, 1 month after surgery, 6 months after surgery, 12 months after surgery, 24 months after surgery and 36 months after surgery
  With this outcome it will be calculated the effect on the quality of life of patients using questionnaire QLQ-CR29.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Arjona Sánchez, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (19):
- Spain (19):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital de Sant Joan Despí. Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitario de Gran Canaria "Dr. Negrín", Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital General Universitario Reina Sofía, Murcia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available.
  Individual parcicipant data that underlie the results reportes in this article, after deidenttification (text, tables, figures and appendices)
  The other documents that will be available: study protocol, Statistical Analysis Plan, Informed Consent Form.
  The data will be available beginning 9 months and ending 36 months following article publication.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: To obtain the data, a proposal must be sent to uicec@imibic.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Arjona-Sanchez A, Espinosa-Redondo E, Gutierrez-Calvo A, Segura-Sampedro JJ, Perez-Viejo E, Concepcion-Martin V, Sanchez-Garcia S, Garcia-Fadrique A, Prieto-Nieto I, Barrios-Sanchez P, Torres-Melero J, Ramirez Faraco M, Prada-Villaverde A, Carrasco-Campos J, Artiles-Armas M, Villarejo-Campos P, Ortega-Perez G, Boldo-Roda E, Sanchez-Hidalgo JM, Casado-Adam A, Rodriguez-Ortiz L, Aranda E, Cano-Osuna MT, Diaz-Lopez C, Romero-Ruiz A, Briceno-Delgado J, Rufian-Pena S; Grupo Espanol de Carcinomatosis Peritoneal. Efficacy and Safety of Intraoperative Hyperthermic Intraperitoneal Chemotherapy for Locally Advanced Colon Cancer: A Phase 3 Randomized Clinical Trial. JAMA Surg. 2023 Jul 1;158(7):683-691. doi: 10.1001/jamasurg.2023.0662. PMID 37099280
- [Derived] Arjona-Sanchez A, Barrios P, Boldo-Roda E, Camps B, Carrasco-Campos J, Concepcion Martin V, Garcia-Fadrique A, Gutierrez-Calvo A, Morales R, Ortega-Perez G, Perez-Viejo E, Prada-Villaverde A, Torres-Melero J, Vicente E, Villarejo-Campos P, Sanchez-Hidalgo JM, Casado-Adam A, Garcia-Martin R, Medina M, Caro T, Villar C, Aranda E, Cano-Osuna MT, Diaz-Lopez C, Torres-Tordera E, Briceno-Delgado FJ, Rufian-Pena S. HIPECT4: multicentre, randomized clinical trial to evaluate safety and efficacy of Hyperthermic intra-peritoneal chemotherapy (HIPEC) with Mitomycin C used during surgery for treatment of locally advanced colorectal carcinoma. BMC Cancer. 2018 Feb 13;18(1):183. doi: 10.1186/s12885-018-4096-0. PMID 29439668